CLINICAL TRIAL: NCT02291926
Title: Phase I Study of Human Umbilical Cord Mesenchymal Stem Cell Implantation in the Treatment of Articular Cartilage Defect of Knee
Brief Title: Human Umbilical Cord Mesenchymal Stem Cell Transplantation in Articular Cartilage Defect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Hornetcorn Bio-technology Company, LTD (Industry)
Collaborators: Fifth Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYK-Articular Cartilage Defect
Record Dates: First submitted 2014-11-07; First posted 2014-11-17 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2015-07

CONDITIONS: Cartilage Diseases; Osteoarthritis
Keywords: Human Umbilical Cord Mesenchymal Stem Cell; Mesenchymal Stem Cell; Osteoarthritis
MeSH Terms: conditions — Cartilage Diseases; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hUC-MSC treatment (Experimental): Patients will receive human umbilical cord mesenchymal stem cells transplantation with a 12 months follow-up.
  Interventions: Biological: Human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cells — A single dose of 2×107 hUC-MSC will be implanted to patients by intra-articular injection, and repeated every month for four times.
  Other Names: hUC-MSC

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of human umbilical cord mesenchymal stem cell(hUC-MSC) for articular cartilage defect of knee.

DETAILED DESCRIPTION:
Human articular cartilage has limited repair potential.Cell-based strategies have explored chondrocytes and mesenchymal stem cells (MSCs) with extensive basic science and preclinical studies.However the concept of autologous chondrocyte implantation is not ideal,so the focus in cartilage repair is shifting toward mesenchymal stem cells.

To investigate the effects of hUC-MSC treatment for articular cartilage defects, 20 patients will be enrolled and receive 4 times of hUC-MSC transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must consent in writing to participate in the study by signing and dating an informed consent document
* Healthy patients with no major history of illness
* Patients must have a diagnosis of osteoarthritis by radiographic criteria of Kellgren and Lawrence grade 2-4
* Patients who needs invasive interventions of arthroplasty due to no response from existing pain medication
* Patients must have had more than Grade 4 (0~10 point numeric scale) pain at least for four months
* Patient's damaged cartilage area should be in the range of 2-6cm2

Exclusion Criteria:

* Pregnant women or lactating mothers
* Patients who have received any anti-inflammatory drugs including herb-drug within 14 days
* Patients who received any drug by intra-articular injection for treatment within 2 months prior to this enrollment
* Patients with positive human immunodeficiency (HIV) at screening indicative of current of pass infection
* Impaired liver function, abnormal blood coagulation, combine other tumor or special condition
* Patients who had participated in other clinical trials within three months prior to this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Severity of adverse events | 12 months
  Adverse events were categorized using National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.0 scale (NCI-CTCAE v4.0).

SECONDARY OUTCOMES:
Magnetic resonance imaging (MRI) of the knee | Before and 1,3,6,12 month after treatment
  The size, depth of cartilage defect, and regenerated cartilage were measured using MRI.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Before and 1,3,6,12 month after treatment
  Change in WOMAC pain score,composite score and function and stiffness index scores.

CONTACTS AND LOCATIONS:
Overall Officials: Ping J Chen, Professor, Principal Investigator — Fifth Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Fifth Affiliated Hospital Immunotherapy center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided